CLINICAL TRIAL: NCT05418478
Title: The Effect of Training Given to Patients With Heart Failure Through Transtheoretic Model-based Telehealth Methods on Self-care, Drug Adherence and Quality of Life
Brief Title: The Effect of Education Given to Patients With Heart Failure on Self-care, Drug Compliance and Quality of Life.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, İbrahim Caner Di̇ki̇ci̇, Lecturer, Harran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 46811200
Record Dates: First submitted 2022-05-31; First posted 2022-06-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: Heart Failure; Transtheoretic model; Treatment Compliance; Self-care; Tele-health; Patient education
MeSH Terms: conditions — Heart Failure; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Intervention Model: Parallel Assignment Masking: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Study group intervention: 7 sessions of transtheoretical model-based interview (2 in the first month, a total of 7 times, once a month), a structured disease education through transtheoretical model-based telehealth practices, and 6-month follow-up.
  * After the participants are included in the study, a health education structured according to the Transtheoretical model will be given to the patients in the study group through tele-health applications.
  * The patients in the intervention group will be trained through tele-health practices for at least 25-30 minutes on a transtheoretical basis, every 2 weeks in the first month and once a month in the following months. Tele-health applications include phone monitoring, SMS notification and application applications.
  * In the 6-month follow-up, there will be 2 follow-ups as pre-test (1st month) and post-test (6th month).
  * Behavioral: 7 sessions of behavior change training based on the transtoerytic model
  Interventions: Behavioral: Intervention transtheoretical model group
- Control (No Intervention): * No notification will be made to the relatives of the patients in the control group. Control group patients will be called for routine control in line with their usual plans. After a total of 6 months from the beginning, the self-care and treatment compliance levels of the patients in the control group will be examined.
  * There will be 2 follow-ups as pre-test (1st month) and post-test (6th month).

INTERVENTIONS:
Behavioral: Intervention transtheoretical model group — The Transtheoretical Model is a conscious behavior modification model that focuses on individual decision making and planning processes. It is the only model that examines behavior change as a dynamic process rather than an outcome, and considers behavioral strategies that include the individual's cognitive and behavioral processes in this process.
  In the model, it is stated that behavior change is a process and develops gradually. It is reported that the change in the behavior of individuals consists of six stages: 1) not thinking, 2) thinking, 3) preparation, 4) taking action, 5) maintaining and 6) terminating. This model consists of four main constructs called change stages (time-related dimension), change processes/behavior modification methods (independent variable dimension), self-efficacy (levels of change) and decision-making balance (perceptions of harm and benefit of change).
  Arms: Intervention group

SUMMARY:
This study was planned as a randomized, controlled, experimental study to evaluate the effects of transtheoretic model-based education on self-care, drug compliance and quality of life in patients with heart failure. The number of samples required for the study was determined by the power analysis made in the GPower 3.1 package program. Assuming that there may be losses in follow-up and considering that non-parametric tests can be performed, the research group will consist of a total of 72 people, 36 in each group, with an increase of 20%. Patients with heart failure who do not have communication barriers to affect cognitive functions, can use tele-health applications (Smartphone and application), volunteers aged 18 and over and agree to participate in the study will be included in the intervention and control groups. The data of the study, "Socio-demographic Characteristic Data Form", "Question Form Regarding the Disease", "European Heart Failure Self-Care Behaviors Scale-12", "Beliefs About Medication Adherence Scale," in which socio-demographic characteristics and information about the disease were questioned. (IUHIO)'' and ''Minnesota Life with Heart Failure Questionnaire''.

DETAILED DESCRIPTION:
The patients in the intervention group will be trained through tele-health practices for at least 25-30 minutes on a transtheoretical basis, every 2 weeks in the 1st month and once a month in the following months. Tele-health applications include phone monitoring, SMS notification and application applications. Educational topics based on model-based self-care behaviors; It will include regular exercise, nutrition-weight monitoring, fluid intake-edema control, smoking cessation, regular drug use, regular rest, vaccination. Educational principles will be shared with patients by SMS from time to time during the education process. Treatment compliance levels and self-care behaviors of both groups of patients will be re-measured from the first week to the 6th month after the training, and any difference will be analyzed using statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Have no communication barriers to affect cognitive functions,
* Ejection-Fraction over 20
* Diagnosed with Heart Failure for at least 6 months
* Able to use tele-health applications (smartphone and application)

Exclusion Criteria:

* Patients with communication difficulties
* Patients who cannot use tele-health applications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
European Heart Failure Self-Care Behaviors Scale | Baseline-6 months
  The scale includes recognizing symptoms such as edema and weight gain, dyspnea, and fatigue associated with heart failure; It consists of 12 questions to measure self-care behaviors such as applying to a doctor and nurse for these symptoms, regular use of drugs, use of fluid and salt, treatment such as diet and exercise regimen and self-care behaviors such as weight monitoring and edema monitoring.

SECONDARY OUTCOMES:
Medication Compliance Notification Scale | Baseline-6 months
  The total test score is obtained by summing the scores obtained from the scale items evaluating drug compliance. Scores from the scale range from 5 to 25. An increase in the obtained scores indicates compatibility, and a decrease in scores indicates inconsistency.
Minnesota Life with Heart Failure Survey | Baseline-6 months
  The scale measures the effect of physical and social functionality on heart failure, as well as assessing the effect of common physical symptoms such as shortness of breath, fatigue, peripheral edema, anxiety and depression symptoms. The 21-item scale is in a six-point Likert type (never=0, very little=1, little=2, a little=3, a lot=4, a lot=5). The lowest score that can be obtained from the scale is 0, and the highest score is 105.
New York Heart Association classification (NYHA) | Baseline-6 months
  Classification of the clinical picture according to the functional status of the patients, from 1 to 4, patients are classified according to their physical activities.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim C Di̇ki̇ci̇, MSc, Study Director — Harran Üniversitesi; Medet Korkmaz, PhD, Study Chair — Inonu University
Locations (1):
- Harran University, Sanliurfa, Türki̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Abbasi A, Ghezeljeh TN, Farahani MA. Effect of the self-management education program on the quality of life in people with chronic heart failure: a randomized controlled trial. Electron Physician. 2018 Jul 25;10(7):7028-7037. doi: 10.19082/7028. eCollection 2018 Jul. PMID 30128093
- [Background] Johnson SS, Paiva AL, Cummins CO, Johnson JL, Dyment SJ, Wright JA, Prochaska JO, Prochaska JM, Sherman K. Transtheoretical model-based multiple behavior intervention for weight management: effectiveness on a population basis. Prev Med. 2008 Mar;46(3):238-46. doi: 10.1016/j.ypmed.2007.09.010. Epub 2007 Oct 23. PMID 18055007
- [Background] Chen H, Wang Y, Liu C, Lu H, Liu N, Yu F, Wan Q, Chen J, Shang S. Benefits of a transtheoretical model-based program on exercise adherence in older adults with knee osteoarthritis: A cluster randomized controlled trial. J Adv Nurs. 2020 Jul;76(7):1765-1779. doi: 10.1111/jan.14363. Epub 2020 May 13. PMID 32202313
- [Result] Lee S, Riegel B. State of the Science in Heart Failure Symptom Perception Research: An Integrative Review. J Cardiovasc Nurs. 2018 May/Jun;33(3):204-210. doi: 10.1097/JCN.0000000000000445. PMID 28858886
- [Result] Paradis V, Cossette S, Frasure-Smith N, Heppell S, Guertin MC. The efficacy of a motivational nursing intervention based on the stages of change on self-care in heart failure patients. J Cardiovasc Nurs. 2010 Mar-Apr;25(2):130-41. doi: 10.1097/JCN.0b013e3181c52497. PMID 20168193
- [Result] Reid KRY, Reid K, Esquivel JH, Thomas SC, Rovnyak V, Hinton I, Campbell C. Using video education to improve outcomes in heart failure. Heart Lung. 2019 Sep-Oct;48(5):386-394. doi: 10.1016/j.hrtlng.2019.05.004. Epub 2019 Jun 4. PMID 31174893
- [Result] Riegel B, Masterson Creber R, Hill J, Chittams J, Hoke L. Effectiveness of Motivational Interviewing in Decreasing Hospital Readmission in Adults With Heart Failure and Multimorbidity. Clin Nurs Res. 2016 Aug;25(4):362-77. doi: 10.1177/1054773815623252. Epub 2016 Jan 6. PMID 26743119